CLINICAL TRIAL: NCT02452398
Title: Clinical Evaluation of Hair Removal and Permanent Hair Reduction for Skin Types V-VI Using Intense Pulsed Light
Brief Title: Clinical Evaluation of Hair Removal and Permanent Hair Reduction for Skin Types VI Using Intense Pulsed Light
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn as technology already proven with data no longer needed.
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0115
Record Dates: First submitted 2015-05-08; First posted 2015-05-22 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Removal of Excess or Unwanted Body Hair
Keywords: Hair removal; depilation; epilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group (Experimental): Hair removal treatment using Venus Versa IPL energy
  Interventions: Device: Treatment group; Other: No intervention
- No intervention (Placebo Comparator): Subject hair count at baseline will act as the control to which the hair count at 6 months after the last treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Treatment group — The intense pulsed light (IPL) applicator with a wavelength of 690 nm and spot size (treatment area) of 30 mm by 10 mm will be used to deliver the energy to the treatment area.
  Arms: Treatment Group
Other: No intervention — Subject will act as their own control where the baseline hair count will be used as a comparator to the hair count after treatment.

SUMMARY:
This is a Multi-center, blinded, baseline-controlled, prospective study to evaluate permanent hair reduction and removal for skin types V and VI using IPL.

DETAILED DESCRIPTION:
One hundred and twenty (120) subjects who are Fitzpatrick Skin Type V-VI, and have a suitable treatment area for hair removal will be evaluated in this study.

Each subject will receive six treatments at four to six week intervals upon re-growth of hair and return for follow-up visits at one, three and six months after the last treatment.

Measurement Equipment Standard High Resolution Digital Camera

Labels for hair count Customized hair count sticker templates will be placed directly on the skin and the hairs in this window will be counted at specific visits during the study as detailed in section.

Study Procedures Each subject will participate in the study for a period of at least 11 months. The study is anticipated to be completed within twelve months.

Test spots Up to 3 test spots will be performed in the selected treatment area to determine the optimal parameters / setting.

Treatment

The treatment areas are divided into 3 groups. Each Subjects will be allocated to one of the following groups::

* Two small anatomical areas (right and left axillae and double sided bikini line) or;
* One double sided large area (right and left thighs) or;
* One large area (whole back / abdomen)

Based on the mild nature of treatment, anesthesia is not required. Before starting treatment apply a layer of conductive gel to the treatment area.

After applying the conductive gel, locate the applicator in close contact, perpendicular to the skin with no pressure applied. Pressing the applicator will fire the IPL pulse. In order to ensure full coverage of the treatment area applicator placement should overlap approximately 1/3 of the previously treated skin.

Post-treatment Instructions Cold packs may be placed on the treated area for post treatment cooling. Subjects should be aware that post treatment erythema, edema and some discomfort of the treated areas are possible and should not be a cause for concern. They may also experience some purpura in the treated areas which would be expected to resolve within several days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written Informed Consent;
2. Subject has black or dark brown terminal hairs in the areas to be treated.
3. Terminal hair density requirement of greater than 15 hairs within the hair count site (3x3 cm area) as determined by manual hair count performed by the study investigator.
4. Healthy adult, male or female, 21 years of age or older with skin type V-VI;
5. Having a suitable treatment area for hair removal;
6. Able and willing to comply with the treatment/follow-up schedule and requirements;
7. Women of child-bearing potential (women who have not had a hysterectomy, bilateral oophorectomy or are not postmenopausal) are required to be using a reliable method of birth control at least three months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Subject has light ,gray terminal or fine hairs in all/some parts of the treated area;
2. Pregnant, expectation of pregnancy, postpartum or nursing (<6 months);
3. Hormonal disorders that may affect hair growth;
4. Immunosuppressive diseases, including AIDS and HIV infection, or use of immunosuppressive medications;
5. Livedo reticularis;
6. Uncontrolled systemic diseases such as diabetes;
7. Active infections in the treated area;
8. Dysplastic nevi;
9. Significant concurrent skin conditions or any inflammatory skin conditions;
10. Active cold sores, open lacerations or abrasions;
11. Chronic or cutaneous viral, fungal, or bacterial diseases;
12. Current cancer;
13. History of skin cancer or pre-cancerous lesions at the treatment areas;
14. Use of Accutane™ (Isotretinoin) within the past six month;
15. Keloid or Hypertrophic scar formation in the treatment area;
16. Tattoos in the treatment area;
17. Bleeding coagulopathies or use of anticoagulants;
18. Auto-immune disorders;
19. Erythema abigne, when identified treatments should be discontinued;
20. Photosensitivity disorder that can be exacerbated by laser or intense light;
21. Herpes simplex in the treatment area;
22. Use of medications, herbal supplements, perfumes or cosmetics that may affect sensitivity to light;
23. Poor wound healing;
24. Sunburns;
25. Unable or unlikely to refrain from artificial tanning, including the use of tanning booths, prior (at least a month) and during the course of the evaluation;
26. Prior skin treatment with laser or other devices on the same treated areas within the last six months prior to study enrollment or during the course of the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2015-01; Primary Completion 2017-03-27 (Actual); Study Completion 2017-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Mancuso, Study Director — Venus Concept
Locations (1):
- Dermatology and Laser Centre, Manhattan Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated and no results analysis was done.
Groups:
- Treatment Group: Hair removal treatment using Venus Versa IPL energy
  Venus Versa: The Venus Versa system is a multi-application device intended to be used in aesthetic and cosmetic procedures.
  The device consists of a console and 4 detachable applicators that deliver optical energy in the form of Intense Pulsed Light to the patient skin. The intense pulsed light lamp delivers light distributed over a range of wavelengths from 500 nm to 1200 nm. Different filters are embedded in the different applicators so that each applicator can deliver the desired spectrum according to the indications to be treated. The applicator that will be used for this study (HR 690) has a wavelength of 690 nm and has a spot size (treatment area) of 30 mm by 10 mm.
  IPL gel: water based gel used to protect the skin during light based treatments. Also used during ultrasound treatments.
Period: Overall Study
Arm/Group | Treatment Group
Started | 79 (Study was halted prematurely. No results analysis completed.)
Completed | 38 (Study was halted prematurely. No results analysis completed.)
Not Completed | 41
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 28
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 6
Not completed — Moved away | 4

BASELINE CHARACTERISTICS:
Population: Data were not collected.
Groups:
- Hair Removal With Versa HR 690nm Applicator: Subjects with Fitzpatrick skin type V-VI requesting hair removal (right and left axillae and double sided bikini line) or one double sided large area (right and left thighs) or one large area (whole back / abdomen).
Arm/Group | Hair Removal With Versa HR 690nm Applicator
Number analyzed (Participants) | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 79
Hair count in marked treatment area [Count of Participants; unit: Participants] — Population: Data were not collected.

OUTCOME MEASURES:

1. Primary Outcome: Hair Count 6 Months Following Last Treatment
Description: Hair count reduction in marked treatment area assessed from photographs taken 6 months following the last treatment as compared to photographs of the marked treatment area taken at baseline.
Time Frame: 6 months after last treatment
Population: This primary outcome measurement could not be reported as data were not collected.
Groups:
- Treatment Group: Enrolled subjects acted as their own control. Each received Venus Versa IPL treatment to remove hair in marked treatment area.
Arm/Group | Treatment Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The adverse event data was collected over a period of 2 years and 2 months.
Groups:
- Hair Removal With Versa HR 690nm Applicator: All subjects who received at least one hair removal treatment with the Versa HR 690 nm applicator.
Arm/Group | Hair Removal With Versa HR 690nm Applicator
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 0/79
Other Adverse Events (participants affected / at risk) | 0/79

LIMITATIONS AND CAVEATS:
The study was terminated due to slow recruitment (over 2 years and the target enrollment had not been reached).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT02452398/Prot_SAP_000.pdf